CLINICAL TRIAL: NCT02235493
Title: A Single-Center, Non-interventional Substudy of ALX-HPP-502 to Assess Functional Natural History Data of Patients With Juvenile Historical Controls in ENB-006-09
Brief Title: Non-interventional Substudy of ALX-HPP-502 to Assess Natural History of Patients With Juvenile-onset HPP Who Served as Historical Controls in ENB-006-09
Status: Completed | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALX-HPP-502s
Record Dates: First submitted 2014-09-05; First posted 2014-09-10 (Estimated); Results first posted 2015-09-28 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Hypophosphatasia; Bone Disease
Keywords: HPP; Soft Bones; low Alkaline Phosphatase; genetic metabolic disorder; alkaline phosphatase; tissue non-specific alkaline phosphatase; rickets; osteomalacia
MeSH Terms: conditions — Hypophosphatasia; Bone Diseases; Rickets; Osteomalacia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Retrospective Case Only
  Interventions: Biological: Retrospective Case Only

INTERVENTIONS:
Biological: Retrospective Case Only

SUMMARY:
The purpose of this study is to characterize the natural history of HPP in patients with Juvenile-onset HPP who served as historical controls in ENB-006-09.

DETAILED DESCRIPTION:
Hypophosphatasia (HPP) is a life-threatening, genetic, and ultra-rare metabolic disease characterized by defective bone mineralization and impaired phosphate and calcium regulation that can lead to progressive damage to multiple vital organs, including destruction and deformity of bones, profound muscle weakness, seizures, impaired renal function, and respiratory failure. There are no approved disease-modifying treatments for patients with this disease. There is also limited data available on the natural course of this disease over time, particularly in patients with the juvenile-onset form.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent/assent prior to video collection and data abstraction.
* Documented informed consent/assent in Study ALX-HPP-502.
* Patients with juvenile-onset HPP and was selected as a historical-control for Study ENB-006-09.
* Patients with at least 2 videos of basic mobility that were recorded at 2 different clinic visits when the patient was ≥5 to ≤15 ye

Exclusion Criteria:

* There are no exclusion criteria for this study

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient has juvenile-onset HPP and was selected as a historical-control for Study ENB-006-09.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2014-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- St Louis, Missouri, United States

REFERENCES:
- See also: Hypophosphatasia Website — http://www.hypophosphatasia.com
- See also: Hypophosphatasia Website for Health Care Professionals — http://www.hypophosphatasia.com/hcp/
- See also: HPP support group — http://www.magicfoundation.org
- See also: US Hypophosphatasia Group (Soft Bones) — http://www.softbones.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Retrospective Observational: Patients diagnosed with juvenile-onset hypophosphatasia (HPP) [ie, documented onset of first signs/symptoms of HPP at ≥ 6 months to < 18 years of age].
Period: Overall Study
Arm/Group | Retrospective Observational
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients who met all of the inclusion and none of the exclusion criteria were defined as the enrolled population, which was also the analysis population.
Arm/Group | Retrospective Observational
Number analyzed (Participants) | 6
Age, Customized [Mean (Standard Deviation); unit: months] — Age at Diagnosis
  months | 28.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race/Ethnicity, Customized [Number; unit: participants]
  White, Hispanic or Latino | 2
  White, Not Hispanic or Latino | 4
Region of Enrollment [Number; unit: participants]
  United States | 6
Modified Performance-Oriented Mobility Assessment - Gait subtest (MPOMA-G) [Median (Inter-Quartile Range); unit: units on a scale] — The MPOMA-G is a 5-component assessment that is used to evaluate gait performance. The first component has 4 sub-components. For 2 components and 2 sub-components, scores of 0 or 1 are assigned while scores of 0, 1 or 2 are assigned to the rest of the 2 components and 2 sub-components based on type of ambulation pattern observed. The maximum total score of 12 points = no impairment and 0 points = worst impairment.
  units on a scale | 6.00 [4.00 to 8.00]
Deceased/Alive Status - Deceased [Number; unit: participants] | 0
Deceased/Alive Status - Alive [Number; unit: participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: Modified Performance-Oriented Mobility Assessment-Gait Subtest (MPOMA-G) - Change From Baseline to Last Overall
Description: The MPOMA-G is a 5-component assessment that is used to evaluate gait performance. The first component has 4 sub-components. For 2 components and 2 sub-components, scores of 0 or 1 are assigned while scores of 0, 1 or 2 are assigned to the rest of the 2 components and 2 sub-components based on type of ambulation pattern observed. The maximum total score of 12 points = no impairment and 0 points = worst impairment.
Time Frame: The earliest available MPOMA-G score that was assessed within the period of patients' aged 5 to 15 years, inclusive.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Retrospective Observational
Number analyzed (Participants) | 6
units on a scale | 1.50 [1.00 to 2.00]
Statistical Analysis 1: Comparison: Retrospective Observational; Videos were reviewed and scored by 3 independent raters who were masked to patient identifiers and the clinic visits and dates when the videos were recorded. Each rater scored the individual components required for the calculation of the total MPOMA-G score for each evaluable patient video. The median of the scores across the 3 raters was obtained for each individual component and summed to generate the median MPOMA-G score used in the analyses; Test type: Superiority or Other; p = 0.0625, Sign test — The p-value is based on a nonparametric sign test to determine whether the median of change from Baseline in MPOMA-G score differs from 0. No multiple comparisons or multiplicity adjustments were conducted

2. Secondary Outcome: Performance-Oriented Mobility Assessment-Gait Subtest (POMA-G) - Change From Baseline to Last Overall
Description: The POMA-G is a 7-component assessment that is used to evaluate gait performance. The second component has 4 sub-components. Scores of 0, 1 or 2 are assigned to 2 components while scores of 0 or 1 are assigned to the rest of the 4 components and 4 sub-components based on type of ambulation pattern observed. The maximum total score of 12 points = no impairment and 0 points = worst impairment.
Time Frame: The earliest available MPOMA-G score that was assessed within the period of patients' aged 5 to 15 years, inclusive.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Retrospective Observational
Number analyzed (Participants) | 6
units on a scale | 1.50 [0.00 to 2.00]
Statistical Analysis 1: Comparison: Retrospective Observational; Videos were reviewed and scored by 3 independent raters who were masked to patient identifiers and the clinic visits and dates when the videos were recorded. Each rater scored the individual components required for the calculation of the total POMA-G score for each evaluable patient video. The median of the scores across the 3 raters was obtained for each individual component and summed to generate the median POMA-G score used in the analyses; Test type: Superiority or Other; p = 0.1250, Sign test — The p-value is based on a nonparametric sign test to determine whether the median of change from Baseline in POMA-G score differs from 0. No multiple comparisons or multiplicity adjustments were conducted

ADVERSE EVENTS:
Time Frame: No adverse event data were collected during this retrospective noninterventional study.
Arm/Group | Retrospective Observational
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Participation in this single-center study involves a commitment to publish the data from the study in a cooperative publication prior to release of study results on an individual basis. Therefore, the PI is subject to certain disclosure and publication limitations.